CLINICAL TRIAL: NCT04009031
Title: Evaluation of a Novel Video Game for Home-based Rehabilitation for Children With Hemiplegic Cerebral Palsy.
Brief Title: Video Game for Home-based Rehabilitation for Children With Hemiplegia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic halted recruitment as of March 2020.
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Brain Institute (Other)
Responsible Party: Principal Investigator, Elaine Biddiss, Doctor, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-365
Record Dates: First submitted 2019-06-14; First posted 2019-07-05 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Child; Hemiplegic Cerebral Palsy
Keywords: video games; upper extremity; rehabilitation; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Participants will undergo a clinical assessment at 3-time points: baseline, post-intervention, and one-month follow-up. Clinical assessments will take approximately 2 hours and will be carried out at the Holland Bloorview Kids Rehabilitation Hospital by an occupational therapist. A research assistant will visit the child's home 3 times throughout the duration of the intervention (weeks 1, 6 and 12). During the last home visit, semi-structured interviews will be conducted individually with the parent and child.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bootle Blast (Experimental): Bootle Blast is a series of 13 mini-games targeting different upper limb motor therapy goals. Bootle Blast is designed with many of the features of mainstream video games known to be appealing to young people. Game rewards are linked to meeting therapeutic objectives, such as daily play targets that are customizable to each child. Bootle Blast is played through movements of the upper limbs tracked via a low-cost camera/sensor (Microsoft Kinect, no hand-held controls needed). The movements required to play are customizable to each child's range of motion. Some of the mini-games are "mixed reality", where children interact and manipulate real-life objects (e.g. musical instruments, coloured building blocks) to play the game. The use of skeletal tracking and mixed reality enables both gross and fine motor skills to be practiced in line with each child's therapy goals and motor abilities.
  Interventions: Device: Bootle Blast

INTERVENTIONS:
Device: Bootle Blast — During the baseline assessment, an occupational therapist will calibrate the video game to the child's therapy needs and functional abilities. Within a week of the first assessment, the research team will set up the video game in the participant's home where it will remain for 12 weeks. Training on how to play the game and a user manual will be provided. The researcher will work with each family to establish a play objective (minutes/day and days/week) that considers the family's schedule. Five-minute telephone check-in calls will be done weekly.

SUMMARY:
This study evaluates the feasibility of a low-cost, movement tracking video game (Bootle Blast) to 1) sustain engagement in children with cerebral palsy (CP) during a 12-week intervention; and 2) generate changes in upper limb functional motor outcomes following the intervention.

DETAILED DESCRIPTION:
Children with Cerebral Palsy (CP) can benefit from home-based practice of therapy exercises. However, sustaining engagement in home-based therapy is challenging. Bootle Blast is a low-cost video game that uses the Microsoft Kinect sensor to track upper limb movements and interactions with real-life objects (e.g. musical instruments, building blocks). To play Bootle Blast, the child needs to use the hemiplegic arm/hand to play unilateral game activities, and highly involve it in bilateral activities.

This study will answer our research questions: 1) to what extent can children achieve a weekly play-time goal (PTG) over a 12-week intervention (adherence) when the PTG is family identified? 2) to what extent can the use of Bootle Blast lead to improvements in UL motor function? and 3) what are the participant's experiences of using BB for home rehabilitation?

As measures of feasibility we hypothesize that 1a) 75% of children will achieve their weekly play time goal and complete the 12-week intervention and 2) 75% children who achieve their weekly play time goal will improve in one or more UL motor outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hemiplegic Cerebral Palsy, Gross Motor Function Classification System and Manual Abilities Classification System Levels I to III, able to co-operate, understand and follow simple instructions for gameplay, live within 30 km of the Holland Bloorview Kids Rehabilitation Hospital, having a caregiver willing to participate.

Exclusion Criteria:

* currently receiving active occupational or physical therapy that may impact motor function of the upper limb, Botulinum Toxin treatment within 3 months or Constraint-Induced Movement Therapy within 6 months of study enrollment, visual, cognitive or auditory limitations at a level that would interfere with gameplay, uncontrolled epilepsy or history of epilepsy related to video game play.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Video game logs | Through out the 12-week intervention.
  Addresses research question 1. Every time the computer is turned on to play the video game, a video game log is automatically generated. The game logs active play time (i.e. time in minutes spent actively engaging in therapeutic movements) and passive play time (e.g. time spent navigating menus). Additional data that is recorded in game logs includes: game scores, games played and time in each game, rewards collected, and location of the joints (e.g. elbow, shoulder) as tracked by the Microsoft Kinect sensor. Data recorded in the video game will be used to identify the percentage of children that met their weekly play time goal, and on how many weeks this goal was achieved.
Change in the Canadian Occupational Performance Measure (COPM) | baseline (week 0), post-intervention (week 13), and follow-up (week 17)
  Addresses research question 2. COPM evaluates self- or parent-reported satisfaction and performance on self-identified therapy goals. Participants will identify, with the help of the occupational therapists during the baseline assessment, 1-3 upper limb goals related to daily life activities (e.g., tie shoelaces). Parent and child will rate together performance and satisfaction with performance on a 10-point scale (1 is poor/low and 10 is good/high) for each goal.
Change in the Assisting Hand Assessment (AHA) | baseline (week 0), post-intervention (week 13), and follow-up (week 17)
  Addresses research question 2. The AHA evaluates the use of the affected hand in assisting during the performance of 22 bimanual activities. Each task is rated on a 4-point rating scale (4=effective, 0= does not do). Tasks include object manipulation from the AHA toy kit, which are scored under the categories of general use, arm use, grasp and release, fine motor adjustments and coordination and pace. Rasch analysis converts raw scores into a logit-based scale ranging from 0-100, with higher scores representing a higher ability.
Semi-structured interviews | Post-intervention (week 13).
  Addresses research question 3. Parent and child will participate in a post intervention semi-structured interview to explore features related to engagement and intervention acceptability.

SECONDARY OUTCOMES:
Change in range of motion | baseline (week 0), post-intervention (week 13) and follow-up (week 17)
  Active range of motion of the shoulder, elbow and wrist will be measured bilaterally via goniometer.
Grip strength | baseline (week 0), post-intervention (week 13) and follow-up (week 17)
  Assesses isometric muscular strength of the hand and forearm. Measured bilaterally via a hand-held dynamometer.
Change in Box and Block test | baseline (week 0), post-intervention (week 13) and follow-up (week 17)
  The test consists a wooden box with two compartments with a vertical division and 150 small cubes. Measures unilateral gross manual dexterity by asking the participant to pass the maximum number of cubes possible above the division, from one side to another, in 60 seconds.
Change in Children's Hand-use Experience Questionnaire (CHEQ) | baseline (week 0), post-intervention (week 13) and follow-up (week 17)
  Captures the child perceived quality and effectiveness of using their affected hand in 29 bilateral tasks. It can be completed by the parent or the child.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Biddiss, PhD, Principal Investigator — Bloorview Research Institute
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Chan-Viquez D, Khan A, Munce S, Fehlings D, Wright FV, Biddiss E. Understanding a videogame home intervention for children with hemiplegia: a mixed methods multi-case study. Front Med Technol. 2023 Jul 12;5:1217797. doi: 10.3389/fmedt.2023.1217797. eCollection 2023. PMID 37502272